CLINICAL TRIAL: NCT03969017
Title: Combination Treatment of Nucleoside （Acid）Analogue (NAs) and Pegylated Interferon α-2b for NAs Treated, Hepatitis B Related, Compensatory Cirrhosis Patients With Low Level Hepatitis b Virus Surface Antigen (HBsAg)
Brief Title: Combination Treatment of NAs and Peg IFN α-2b for Hepatitis B Related, Compensatory Cirrhosis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-CURE VI STUDY
Record Dates: First submitted 2019-05-21; First posted 2019-05-31 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Cirrhosis of Liver Due to Hepatitis B (Disorder)
MeSH Terms: interventions — nas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAs+Peg IFN Group (Experimental): NAs+Peg IFN Group will receive the treatment of NAs (patients previously treated with telbivudine will be changed to entecavir) plus pegylated interferon (Peg IFN)α-2b.
  Interventions: Drug: pegylated interferon (Peg IFN)α-2b; Drug: Nucleoside （acid）analogue (NAs)
- NAs Group (Other): NAs Group will be treated with NAs as before enrollment.
  Interventions: Drug: Nucleoside （acid）analogue (NAs)

INTERVENTIONS:
Drug: pegylated interferon (Peg IFN)α-2b — Participants in NAs+Peg IFN Group will be treated by Peg IFNα-2b （180ug per week, the dose will be changed to 135ug or 90ug per week during the treatment if patients could not tolerate the side effects of Peg IFNα-2b). Peg IFNα-2b treatment will be performed until HBsAg <0.05IU/ml, with a maximum duration of 48 weeks.
  Other Names: Pi Gebin
  Arms: NAs+Peg IFN Group
Drug: Nucleoside （acid）analogue (NAs) — Both of NAs Group and NAs+Peg IFN Group will be treated with NAs as before enrollment.
  Other Names: Boludine

SUMMARY:
The study aims to demonstrate that whether treatment of nucleoside （acid）analogues (NAs) plus pegylated interferon (Peg IFN) α-2b for those NAs treated, low level of HBsAg, hepatitis B related compensatory cirrhosis patients will result in higher HBsAg clearance rate and reduce the risk of liver cancer. The investigators plan to enroll about 84 hepatitis B related compensatory cirrhosis patients, who have received NAs treatment more than 1 year with the level of HBsAg <1000IU/ml. These participants will be devided into 2 groups. Group A will receive the treatment of NAs plus Peg IFNα-2b. Group B will be treated with NAs as before enrollment. The participants in both groups will be followed up for 96 weeks.

The primary endpoint is to compare the clearance rate of HBsAg between two groups. The secondary endpoint includes: (1) comparing the incidence of liver cancer during the 96 weeks follow-up, (2) comparing adverse side effects between the 2 groups. (3) comparing the virological and biochemical responses between the 2 groups.

DETAILED DESCRIPTION:
Clearance of hepatitis B virus surface antigen (HBsAg) is considered to be the ultimate therapeutic goal for hepatitis B patients, for it is related with low incidence of fibrosis and liver cancer. The investigators' previous study show that nucleoside （acid）analogues (NAs) treated, non-cirrhosis hepatitis B patients switched to /or combined with pegylated interferon (Peg IFN)α-2b could obtain a higher HBsAg clearance rate. Hence, the investigators' hypothesis is that treatment of NAs plus Peg IFNα-2b for those NAs treated, low level of HBsAg, hepatitis B related compensatory cirrhosis patients result in higher HBsAg clearance rate and reduce the risk of liver cancer.

The investigators plan to enroll about 84 hepatitis B related compensatory cirrhosis patients, who have received NAs treatment more than 1 year with the level of HBsAg <1000IU/ml. These participants will be devided into 2 groups according to their wishes. Group A will receive the treatment of NAs (patients previously treated with telbivudine will be changed to entecavir) plus Peg IFNα-2b （180ug per week, the dose will be changed to 135ug or 90ug per week during the treatment if patients could not tolerate the side effects of Peg IFNα-2b）. Peg IFNα-2b treatment will be performed until HBsAg <0.05IU/ml, with a maximum duration of 48 weeks. Group B will be treated with NAs as before enrollment. The participants in both groups will be followed up for 96 weeks.

The primary endpoint is to compare the clearance rate of HBsAg between two groups. The secondary endpoint includes: (1) comparing the incidence of liver cancer during the 96 weeks follow-up, (2) comparing adverse side effects, such as ascites, gastrointestinal bleeding, encephalopathy, hepatorenal syndrome between the 2 groups. (3) comparing the virological and biochemical responses between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-65 years old; Clinical diagnosis of compensatory cirrhosis; Child-Pugh grade A; Positive serum hepatitis B surface antigen (HBsAg); HBsAg titer < 1000IU/ml; Treated by nucleoside （acid）analogues (NAs) more than 1 year; HBV DNA <20 IU/ml; Negative serum hepatitis B e antigen (HBeAg); 15 minutes retention rate of indocyanine green <10%; The blood routine examination: 4×10e9/L<WBC<10×10e9/L、100×10e9/L<PLT<300×10e9/L.

Exclusion Criteria:

* Treated by interferon within half a year; Drug induce liver diseases; Autoimmune liver diseases; Liver diseases caused by metabolic factors; Superinfection with hepatitis A, C, D, E viruses; Infected by HIV virus; Severe respiratory diseases; Severe circulatory diseases, ; Severe digestive diseases; Severe neurological diseases; Need for immunosuppressive therapy for other diseases; Need for radiotherapy/chemotherapy for other diseases; Thyroid diseases; Rheumatic diseases; Malignant tumors; Severe varicose esophageal and gastric fundus veins; Mental or psychological disorders; Alcohol or drug abusers (average alcohol consumption >40g/d for men, >20g/d for women); With contraindications to interferon therapy; Pregnancy or having pregnancy plan in 3 years; Lactation; Can not comply with the study protocol; Fail to sign the informed consent; Other conditions that are not suitable for enrollment determined by researchers.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
The clearance rate of HBsAg for both groups during 96 weeks. | 96 weeks
  The clearance rate of HBsAg will be compared between 2 groups.

SECONDARY OUTCOMES:
The incidence rate of liver cancer for both groups during 96 weeks | 96 weeks
  The incidence of liver cancer will be compared between 2 groups.
Occurance rate of adverse side effects in both groups | 96 weeks
  Adverse side effects, such as ascites, gastrointestinal bleeding, encephalopathy, hepatorenal syndrome will be compared between 2 groups
The change of liver functions in both groups | 96 weeks
  The levels of alanine transaminase, glutamic-oxalacetic transaminase, albumin, total bilirubin, INR will be compared between the 2 groups.
The change of blood routine test indexes in both groups | 96 weeks
  The levels of WBC, Hb, PLT will be compared between the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bingliang Lin, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fattovich G, Bortolotti F, Donato F. Natural history of chronic hepatitis B: special emphasis on disease progression and prognostic factors. J Hepatol. 2008 Feb;48(2):335-52. doi: 10.1016/j.jhep.2007.11.011. Epub 2007 Dec 4. PMID 18096267
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B. Hepatology. 2007 Feb;45(2):507-39. doi: 10.1002/hep.21513. No abstract available. PMID 17256718
- [Background] Liaw YF, Chu CM. Hepatitis B virus infection. Lancet. 2009 Feb 14;373(9663):582-92. doi: 10.1016/S0140-6736(09)60207-5. PMID 19217993
- [Background] Thompson AJ, Nguyen T, Iser D, Ayres A, Jackson K, Littlejohn M, Slavin J, Bowden S, Gane EJ, Abbott W, Lau GK, Lewin SR, Visvanathan K, Desmond PV, Locarnini SA. Serum hepatitis B surface antigen and hepatitis B e antigen titers: disease phase influences correlation with viral load and intrahepatic hepatitis B virus markers. Hepatology. 2010 Jun;51(6):1933-44. doi: 10.1002/hep.23571. PMID 20512987
- [Background] Nguyen T, Thompson AJ, Bowden S, Croagh C, Bell S, Desmond PV, Levy M, Locarnini SA. Hepatitis B surface antigen levels during the natural history of chronic hepatitis B: a perspective on Asia. J Hepatol. 2010 Apr;52(4):508-13. doi: 10.1016/j.jhep.2010.01.007. Epub 2010 Feb 16. PMID 20206400
- [Background] Liu J, Lee MH, Batrla-Utermann R, Jen CL, Iloeje UH, Lu SN, Wang LY, You SL, Hsiao CK, Yang HI, Chen CJ. A predictive scoring system for the seroclearance of HBsAg in HBeAg-seronegative chronic hepatitis B patients with genotype B or C infection. J Hepatol. 2013 May;58(5):853-60. doi: 10.1016/j.jhep.2012.12.006. Epub 2012 Dec 13. PMID 23246508
- [Background] Tseng TC, Liu CJ, Su TH, Wang CC, Chen CL, Chen PJ, Chen DS, Kao JH. Serum hepatitis B surface antigen levels predict surface antigen loss in hepatitis B e antigen seroconverters. Gastroenterology. 2011 Aug;141(2):517-25, 525.e1-2. doi: 10.1053/j.gastro.2011.04.046. Epub 2011 Apr 28. PMID 21672542
- [Background] Chang TT, Gish RG, de Man R, Gadano A, Sollano J, Chao YC, Lok AS, Han KH, Goodman Z, Zhu J, Cross A, DeHertogh D, Wilber R, Colonno R, Apelian D; BEHoLD AI463022 Study Group. A comparison of entecavir and lamivudine for HBeAg-positive chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1001-10. doi: 10.1056/NEJMoa051285. PMID 16525137
- [Background] Hou JL, Gao ZL, Xie Q, Zhang JM, Sheng JF, Cheng J, Chen CW, Mao Q, Zhao W, Ren H, Tan DM, Niu JQ, Chen SJ, Pan C, Tang H, Wang H, Mao YM, Jia JD, Ning Q, Xu M, Wu SM, Li J, Zhang XX, Ji Y, Dong J, Li J. Tenofovir disoproxil fumarate vs adefovir dipivoxil in Chinese patients with chronic hepatitis B after 48 weeks: a randomized controlled trial. J Viral Hepat. 2015 Feb;22(2):85-93. doi: 10.1111/jvh.12313. Epub 2014 Sep 22. PMID 25243325
- [Background] Moucari R, Korevaar A, Lada O, Martinot-Peignoux M, Boyer N, Mackiewicz V, Dauvergne A, Cardoso AC, Asselah T, Nicolas-Chanoine MH, Vidaud M, Valla D, Bedossa P, Marcellin P. High rates of HBsAg seroconversion in HBeAg-positive chronic hepatitis B patients responding to interferon: a long-term follow-up study. J Hepatol. 2009 Jun;50(6):1084-92. doi: 10.1016/j.jhep.2009.01.016. Epub 2009 Mar 9. PMID 19376603
- [Background] Dietary effects on diurnal variation in lipogenesis. Nutr Rev. 1987 May;45(5):157-8. doi: 10.1111/j.1753-4887.1987.tb06353.x. No abstract available. PMID 3601258
- [Background] Chevaliez S, Hezode C, Bahrami S, Grare M, Pawlotsky JM. Long-term hepatitis B surface antigen (HBsAg) kinetics during nucleoside/nucleotide analogue therapy: finite treatment duration unlikely. J Hepatol. 2013 Apr;58(4):676-83. doi: 10.1016/j.jhep.2012.11.039. Epub 2012 Dec 3. PMID 23219442
- [Background] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Background] Buster EH, Flink HJ, Cakaloglu Y, Simon K, Trojan J, Tabak F, So TM, Feinman SV, Mach T, Akarca US, Schutten M, Tielemans W, van Vuuren AJ, Hansen BE, Janssen HL. Sustained HBeAg and HBsAg loss after long-term follow-up of HBeAg-positive patients treated with peginterferon alpha-2b. Gastroenterology. 2008 Aug;135(2):459-67. doi: 10.1053/j.gastro.2008.05.031. Epub 2008 May 15. PMID 18585385
- [Background] Moucari R, Boyer N, Ripault MP, Castelnau C, Mackiewicz V, Dauvergne A, Valla D, Vidaud M, Chanoine MH, Marcellin P. Sequential therapy with adefovir dipivoxil and pegylated interferon alfa-2a for HBeAg-negative patients. J Viral Hepat. 2011 Aug;18(8):580-6. doi: 10.1111/j.1365-2893.2010.01332.x. Epub 2010 May 17. PMID 20487260
- [Background] Sarin SK, Kumar M, Kumar R, Kazim SN, Guptan RC, Sakhuja P, Sharma BC. Higher efficacy of sequential therapy with interferon-alpha and lamivudine combination compared to lamivudine monotherapy in HBeAg positive chronic hepatitis B patients. Am J Gastroenterol. 2005 Nov;100(11):2463-71. doi: 10.1111/j.1572-0241.2005.00247.x. PMID 16279901
- [Background] Ning Q, Han M, Sun Y, Jiang J, Tan D, Hou J, Tang H, Sheng J, Zhao M. Switching from entecavir to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: a randomised open-label trial (OSST trial). J Hepatol. 2014 Oct;61(4):777-84. doi: 10.1016/j.jhep.2014.05.044. Epub 2014 Jun 7. PMID 24915612
- [Background] Fattovich G, Giustina G, Realdi G, Corrocher R, Schalm SW. Long-term outcome of hepatitis B e antigen-positive patients with compensated cirrhosis treated with interferon alfa. European Concerted Action on Viral Hepatitis (EUROHEP). Hepatology. 1997 Nov;26(5):1338-42. doi: 10.1002/hep.510260536. PMID 9362381
- [Background] Ikeda K, Kobayashi M, Saitoh S, Someya T, Hosaka T, Akuta N, Suzuki Y, Suzuki F, Tsubota A, Arase Y, Kumada H. Significance of hepatitis B virus DNA clearance and early prediction of hepatocellular carcinogenesis in patients with cirrhosis undergoing interferon therapy: long-term follow up of a pilot study. J Gastroenterol Hepatol. 2005 Jan;20(1):95-102. doi: 10.1111/j.1440-1746.2004.03527.x. PMID 15610453